CLINICAL TRIAL: NCT04212676
Title: The Effect of Body Awareness Therapy on Postural Stability, Balance and Fear of Falling in Patients With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2019.1031
Record Dates: First submitted 2019-12-19; First posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-02

CONDITIONS: Asthma
Keywords: Asthma; Body Awareness Treatment; Postural Stability; Balance; Fear of Falling
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: The type of study is experimental. A computer-based randomization program (random.org) will be used to identify patients to be assigned to the experimental and control groups. All patients in the experimental and control groups will receive a 30-minute Pulmonary Rehabilitation (PR) program every day of the week for 8 weeks. In addition to the PR program, the BAQ will be administered to the experimental group by the physiotherapist. At the end of the eight weeks, all initial assessments will be repeated. All patients will be supervised physiotherapy sessions for 8 weeks and checked how they implement the program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PR+BAT Group (Experimental): In addition to the PR program, the BAT will be administered to the experimental group by a physiotherapist with 5 years of experience in BAT for 8 weeks.
  Interventions: Other: Body Awareness Therapy; Other: Pulmonary Rehabilitation
- PR Group (Active Comparator): Patients in the control groups will receive a 30-minute Pulmonary Rehabilitation (PR) program every day of the week for 8 weeks.
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Body Awareness Therapy — The BAT for the participants was based on the works of Roxendal and Dropsy. Activities include relaxation exercises, breathing exercises, floor exercises for trunk and pelvic movements, weight transfer using extremities and proprioceptive movements. Movements will be made in various positions to determine the centerline of the body. All exercises will be started in the supine position to maximize proprioceptive motion feedback and minimize energy requirements during tasks. Movements will be taught in a series of lessons over a period of 8 weeks with advance advancement of selected movements depending on participant comfort.
  Other Names: BAT
  Arms: PR+BAT Group
Other: Pulmonary Rehabilitation — Diaphragmatic breathing exercise Thoracic expansion exercises (Chest breathing and bilateral segmental breathing exercises) Inductive spirometry (Triflo®) exercise Cough development techniques
  Other Names: PR

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is one of the serious diseases with a high prevalence and mortality, which adversely affects the quality of life, and is expected to rank third in the global burden of disease in 2020. Although the primary pathophysiology of the disease is pulmonary, it is emphasized that extrapulmonary involvement and comorbid conditions adversely affect the severity and prognosis of the disease. In the treatment guidelines for COPD, extrapulmonary systems and symptoms should also be evaluated. In this context, the number of studies on the effects of postural stability, balance and fall has increased recently, especially in COPD patients. Although the efficacy of pulmonary rehabilitation (PR) in COPD is well defined, it provides minimal gains in postural control and balance. Alternative therapies are needed to improve postural stability, balance and fall in COPD patients.

Body Awareness Therapy (BAQ) is an alternative method developed by French exercise instructor and psychotherapist Jacques Dropsy in the early 1970s following the emergence of the concept of body awareness, adapted to rehabilitation programs by Swedish and Norwegian physiotherapists. Traditional physiotherapy methods are the basis of BAQ. In the treatment, sensory stimulation and movement quality, rhythm, coordination, breathing, relaxation, balance, coordination and proprioceptive exercises give more space. In the literature, BAQ decreases pain, fatigue, eating and sleep problems in chronic musculoskeletal or rheumatic pain, coronary artery disease and neurological patient groups. It is seen to increase the quality of exercise, coordination, balance, postural control, quality of life and the integration between mind-body. Movement awareness and mind-body-behavior interaction developed in BAQ can help regulate emotional, mental, social and behavioral factors that affect health. In addition to improving coping skills and cognitive behaviors among COPD patients, it can contribute to positive gains in better movement, respiratory control and balance. The aim of this study is to investigate the effect of BAQ, which is integrated into 8-week pulmonary rehabilitation sessions, on postural stability, balance and fall conditions.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a common disease that can be prevented and treated, usually characterized by persistent respiratory symptoms and airway restriction due to airway and / or alveolar abnormalities due to exposure to harmful particles or gases. At the same time, it was emphasized that COPD is a systemic disease according to GOLD (Global Initiative for Obstructive Lung Diseases) and extrapulmonary involvement and comorbid conditions adversely affect the severity and prognosis of the disease. COPD is a chronic condition in which physical function, social function and general health are severely affected. Treatment in COPD is mainly aimed at effective disease management, prevention of disease progression, improvement of symptoms, and improvement of exercise tolerance. In the treatment guidelines for chronic lung diseases, extrapulmonary systems and symptoms should also be evaluated. In this context, the number of studies on the effects of postural stability, balance and fall has increased recently, especially in COPD patients. It is reported that the ability of the trunk to participate in postural stability due to increased resting breathing load, weakness of the muscle strength of the diaphragm, one of the major muscles with significant impact on balance, weakness of peripheral muscle and systemic inflammation lead to postural stability and balance risk in COPD patients. Clinical investigations of COPD patients in proportion to the severity of the disease; functional balance, coordination and mobility. Postural stability is defined as the act of maintaining, obtaining or recovering an equilibrium state during any posture or activity. Loss of postural control is one of the most common comorbidities in elderly individuals. Impaired postural control is more common when the elderly person has a chronic disease. The PLATINO study showed an increased prevalence of COPD in elderly individuals. Factors such as lower extremity muscle weakness, functional performance deficit and adaptive capacity, and reduced physical activity level in the elderly with COPD affect postural stability. In individuals with COPD, responses to postural perturbations have been shown to decrease compared to healthy controls. However, the ability to produce a successful postural reaction depends not only on motor performance but also on the efficient use of proprioceptive inputs. In a comprehensive study characterizing proprioceptive postural control in COPD, patients concluded that postural stabilization was impaired compared to healthy controls using ankle muscle proprioceptive signals more and back muscle proprioceptive signals less during balance control. These findings may be a potential risk factor for the likelihood of falls in COPD patients. Among the problems associated with COPD, there is considerable evidence that the risk of falls in these individuals increases. Falling problems and COPD are two major problems that bring great costs to the health system and especially affect elderly people. The well-known fall risk factors in COPD patients are lower limb muscle weakness and loss of mobility, characterized by a decrease in daily living activities. Although the efficacy of pulmonary rehabilitation (PR) in COPD is well defined, it provides minimal gains in postural control and balance. Alternative treatments are needed to improve balance and fall in COPD patients.

Body Awareness Therapy (BAT) is an alternative method developed by French exercise instructor and psychotherapist Jacques Dropsy in the early 1970s following the emergence of the concept of body awareness and adapted to rehabilitation programs by Swedish and Norwegian physiotherapists. Traditional physiotherapy methods are the basis of BAT. Focusing on the senses, proprioceptive exercises aiming to improve the quality of movement, rhythm and coordination with sensory stimuli. BAT treats the individual physically, physiologically, psychologically and socially with a holistic approach and the treatment program is shaped according to the patient's needs. Breathing exercises, relaxation exercises, movement approaches specific to sensory awareness, positioning, stabilization, improving rhythm and coordination, and improving the ability to perform the exercise with maximum awareness are used in physiotherapy methods used in BAT. It consists of specific exercises, which include focusing on how the body is used during movements, aiming at improving one's awareness, ability to be careful, and quality of movement. In the literature, it is seen that Body Awareness Therapy reduces pain, fatigue, eating and sleep problems in various patient groups and increases the quality, coordination, balance, postural control, quality of life and mind-body integration of the exercise.

VFT has been gaining popularity in recent years among many health professionals, especially physiotherapists. In BAT, movement is expressed by how one copes with the balance of the person and associates himself / herself with the place and vertical axis in relation to the environment. The integrity of postural stability is essential for comfortable breathing and awareness, key points for dynamic balance, and quality of movement. Although VFT consists of simple repetitive movements that maintain the ability to use stability limits, its main component is to increase the individual's awareness of his / her movements. Thanks to the neuroplasticity of the brain; multiple slow repetitive movements allow the participant to experience the body and its limits. Movement consciousness that develops by cortical processing of information about movement in the brain and facilitation of proprioceptive; postural control improves balance and coordination. In many cases that require treatment as a principled movement training technique behind mind-body interaction, which emphasizes motion teaching based on sensory motor awareness and cognitive perception of movement. BAT aims to normalize posture, balance, muscular tension and stiffness. Experiences learned by patients help them divide difficult movements into simpler, lighter movements with less energy consumption. Movement awareness and mind-body interaction during movement therapy can help regulate emotional, mental, social and behavioral factors that affect health. In addition to improving coping skills and cognitive behaviors among COPD patients, investigators think that integrating them into pulmonary rehabilitation sessions can have positive effects on postural stability, balance and fall, as they can help them move better and help postural control and thus improve their ability to perform daily living activities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD according to GOLD and willingness to participate
* Age between 40-80 years
* Clinically stable period
* No serious hearing and vision problems

Exclusion Criteria:

* Patients with recurrent exacerbations reported (history of exacerbation in the last two months)
* Having cognitive impairment (less than 24 Mini Mental Test scores)
* Having diagnosed vision, hearing, vestibular or neurological problems that may affect balance
* Having diagnosed orthopedic problems affecting mobility or having a history of surgical intervention
* COPD patients receiving home oxygen therapy or frequent need of oxygen therapy
* Patients with exercise-induced dyspnea
* Patients with primary pulmonary hypertension or patients with pulmonary embolism
* Congestive heart failure and severe coronary patients with coronary artery disease or by-pass surgery due to coronary artery disease
* Patients with morbid obesity
* Presence of systemic disease involving the lung and lung that would previously cause dyspnea other than COPD
* Having received pulmonary rehabilitation in the last 12 months
* Presence of unstable cardiovascular disease
* SpO2<90%
* Problems with understanding and co-operation in understanding tests

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Postural Stability | 8 weeks
  In our study, the postural stability levels of the cases will be evaluated with their feet wide open on the balance platform without any support. The subjects were asked to hold the ball at the midpoint of the circle on the screen opposite to the position and center of gravity of the individual and to keep it at the midpoint for 1 minute; During the measurement, right - left and anterior - posterior oscillations and overall performance levels of the subjects will be recorded.
Balance | 8 weeks
  Balance Master device will be used. Using a fixed 18 "x 60" force platform, the Balance Master determines the vertical force exerted by the patient's feet to measure the center of balance.
Fear of Falling | 8 weeks
  It will be evaluated by the Drop Efficacy Scale. ISI is a 10-item scale. They are asked to score between 1 and 10 to the questions. 1 means a lot of trust, 10 means no. A total score of 0 to 100 is obtained. If the total score is more than 70 points, there is fear of falling.

SECONDARY OUTCOMES:
Tiffeneau index for Pulmonary Function Test | 8 weeks
  Tiffeneau index, also called FEV1 / FVC ratio will be used. FEV1 / FVC ratio is defined as obstruction if less than 70% and restriction if more than 80%.
The Medical Research Council Dyspnea Scale (mMRC) for dyspnea | 8 weeks
  The Medical Research Council Dyspnea Scale (mMRC) use to determine the degree of dyspnea on daily activities. The mMRC dyspnea scale determines the risk of future mortality and includes five dyspnea questions. The scale is scored between 0-4 degrees. Increased grade means severe dyspnea.
6-Minute Walk Test (6MWT) for functional capacity | 8 weeks
  The distance traveled by the subjects as fast as possible at their own walking speed for 6 minutes in a 30-meter straight corridor, but without running will be recorded in meters. The elongation of the distance indicates an increase in the functional capacity of the patient.
Chronic Obstructive Pulmonary Disease Assessment Test (CAT) | 8 weeks
  Chronic Obstructive Pulmonary Disease Assessment Test (CAT): An eight-item, short, easy-to-use clinical test that evaluates the effects of COPD (cough, sputum, fatigue, confidence in leaving home) and deterioration in the patient's health. Scores range from 0-40. The higher the score, the higher the severity of the disease.
Self-Efficacy Scale for the assessment of disease compliance: | 8 weeks
  Assessment of Disease Compliance will be evaluated by the Self-Efficacy Scale in Chronic Diseases. It was developed by Lorig et al. (1996) to measure self-efficacy perceptions of individuals with chronic disease. The scale consists of three main concepts and a total of 10 sub-dimensions. The scale is answered in likert type which determines the self-efficacy perception increasing from 1 to 10. Number 1 in the scale represents yok I have no confidence, and number 10 represents "I have full confidence". The total score of the individual is divided by the number of items and an average self-efficacy score is found. If this score is below 7, it means that strategies and problem-solving must be reassessed to prevent failure. A score of 7 or higher means that the individual has high self-efficacy and can achieve his / her thoughts. a minimum of 10 and a maximum of 100 points can be obtained from the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Karaca, MsC, Principal Investigator — Marmara University; Aysel Yıldız Özer, Ass.Prof.Dr., Study Chair — Marmara University; Sait Karakurt, Prof. Dr., Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karaca S, Yildiz Ozer A, Karakurt S, Polat MG. Effects of body awareness therapy on balance and fear of falling in patients with chronic obstructive pulmonary disease: a randomized controlled trial. Biopsychosoc Med. 2024 Feb 26;18(1):6. doi: 10.1186/s13030-024-00303-x. PMID 38409129